CLINICAL TRIAL: NCT03664869
Title: Intravesical Instillation Therapy With Bacillus Calmette-Guérin (BCG) and Sequential BCG and Electromotive Mitomycin-C (EMDA-MCC) in Patients With High-risk Non-muscle-invasive Bladder Carcinoma
Brief Title: Electromotive Mitomycin-C (EMDA-MMC) in Preventing Recurrences in High-risk Non-muscle-invasive Bladder Cancer
Acronym: FB10
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Finnbladder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Finnbladder-10
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; recurrence; BCG; mitomycin C; electromotive drug administration
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence | interventions — BCG Vaccine; BCG Connaught

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): BCG instillation therapy with induction period of six weekly instillations of BCG followed by maintenance period of ten monthly instillations of BCG
  Dosage of Bacillus of Calmette-Guerin (BCG) is dependent on the preferred brand of BCG by the participating institution. Either 2 x 10^8 - 3 x 10^9 for BCG-MEDAC, 2-8 x 10^8 colony forming unit for OncoTICE or, 81mg for ImmuCYST and TheraCys. The investigators will nominate which BCG brand is used.
  Interventions: Drug: BCG instillation therapy
- Group B (Experimental): Sequential BCG and EMDA mitomycin C treatment with nine weekly instillations of BCG, BCG, EMDA-MMC x3 followed by nine monthly instillations of EMDA-MMC, EMDA-MMC, BCG x3
  Dosage of Bacillus of Calmette-Guerin (BCG) is dependent on the preferred brand of BCG by the participating institution. Either 2 x 10^8 - 3 x 10^9 for BCG-MEDAC, 2-8 x 10^8 colony forming unit for OncoTICE or, 81mg for ImmuCYST and TheraCys. The investigators will nominate which BCG brand is used.
  Mitomycin C dosage is 40 mg of MMC with 960 mg of excipient sodium chloride dissolved in 100 ml sterile water
  Interventions: Drug: Sequential BCG and EMDA mitomycin C

INTERVENTIONS:
Drug: BCG instillation therapy — Induction period of six weekly instillations of BCG followed by maintenance period of ten monthly instillations of BCG
  Other Names: BCG; BCG-MEDAC; OncoTICE; ImmuCyst; TheraCys
  Arms: Group A
Drug: Sequential BCG and EMDA mitomycin C — Induction period includes nine weekly instillations of sequential BCG and EMDA-MMC instillations applied as three cycles of BCG, BCG and EMDA-MMC. Induction period is followed by maintenance period of nine monthly instillations of sequential EMDA-MMC and BCG applied with three cycles of EMDA-MMC, EMDA-MMC and BCG.
  BCG instillation is performed as a standard instillation.
  Mitomycin C is administered with electromotive drug administration (EMDA) device (Instillation: 40 mg mitomycin C with 960 mg of excipient sodium chloride dissolved in 100 ml sterile water, EMDA settings: current rise rate 30-50 microamperes per second, max 25 milliamperes, treatment duration 30 min)
  Other Names: Sequential BCG and EMDA-MMC
  Arms: Group B

SUMMARY:
Disease recurrence and progression is a major issue in high risk non-muscle-invasive bladder cancer (NMIBC).

The current study compares two adjuvant instillation therapies in the treatment of high risk NMIBC. After resection of the tumour(s), patients will receive either traditional regimen of Bacillus Calmette-Guérin (BCG) instillations or combination treatment consisting of sequential BCG-instillations and mitomycin C instillations administered with electromotive drug administration (EMDA) device.

DETAILED DESCRIPTION:
Non-muscle-invasive bladder cancer (NMIBC) is a heterogeneous disease. The patients with NMIBC may be categorized in three risk groups according to the risk of recurrence and progression characterized by the disease. The treatment of high risk NMIBC includes a transurethral resection of the tumour(s), which is followed by an adjuvant instillation therapy, aiming to reduce the risk of recurrence and progression. Intravesical bacillus Calmette-Guérin (BCG) treatment is been the most effective single agent against NMIBC, and it is referred to as the gold standard in the treatment of high risk disease.

BCG is a solution of live, attenuated mycobacterium bovis bacteria, which is administered intravesically in an outpatient clinic. BCG activates an immunological reaction in the bladder wall, which leads to antitumour effect by activation of macrophages, T-cells, and natural killer (NK) cells. BCG treatment comprises an induction period, which includes six weekly instillations. This is followed by maintenance period including monthly or repeated series of three weekly instillations up to 1-3 years.

Other instillation therapies include intravesically administered chemotherapy. Mitomycin C (MMC) is the most used chemotherapeutic agent. MMC provides a better tolerated side effect profile, but is less effective against high risk NMIBC than BCG, when MMC is used as a single agent. Combinations of BCG- and MMC treatment has also been described with various results. The rationale for combining BCG and MMC is to enhance the absorption of BCG as MMC might cause disruption of bladder mucosa, which makes the mucosa more permeable thus enhancing the absorption of BCG. However, it is also hypothesized, that BCG may also work synergistic in favor of MMC.

The absorption and effect of MMC may be enhanced with electromotive drug administration (EMDA) device. After instillation of MMC, an electric field is conducted in the bladder with EMDA device via catheter and electrodes, which are placed in the bladder and lower abdomen skin. Electric field creates movement of sodium ions and water into the bladder wall, which creates electro-osmotic drag of MMC molecules. In a laboratory setting, EMDA-MMC instillation results in 4-7 times greater concentration of MMC in the deeper layers of the bladder wall than passively administered MMC instillation. EMDA-MMC treatment may also be combined with BCG treatment administering BCG and EMDA-MMC instillations sequentially. Results from a prospective randomized trial suggested, that sequential EMDA-MMC and BCG treatment might be even more effective against NMIBC than BCG therapy alone in terms of recurrence, progression and overall survival.

The current study is a prospective, open label, phase III randomized study allocating patients with high risk NMIBC to receive adjuvant instillation therapy either as traditional BCG treatment, or sequential BCG- and EMDA-MMC treatment. The aim of the study is to compare effectiveness and tolerability of the two treatment regimens in preventing recurrence and progression of high risk NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-muscle-invasive tumour types confined to the urinary bladder
* Carcinoma in situ with or without a papillary tumour(s)
* Ta tumour(s) of high-grade
* Any T1 tumour(s)
* Written informed consent is required from every eligible patient
* Second resection performed in case of T1 tumour
* Adequate physical and mental condition to participate in the study (as judged by treating physician

Exclusion Criteria:

* Ta low grade tumour(s)
* Muscle invasive (pT≥2) tumors
* Urothelial cancer involving the prostatic urethra or upper urinary tract
* Non-urothelial bladder cancer.
* Prior BCG failure (If the patient has previously been successfully treated with BCG, and duration from the last instillation is >12 months, participation may be considered, if bladder preserving is chosen)
* Prior or concurrent immunotherapy
* Any medication or condition considered as contraindication to BCG or MMC (as judged by the treating physician)
* Urethral stricture, stone disease, chronic urinary tract infection or any other urological condition that may comprise study participation (as judged by the treating physician)
* Known allergy to MMC or BCG
* Age < 18 years
* Pregnancy or lactating patient
* Other untreated or unstable malignancy in risk of recurrence/progression (as judged by the treating physician)
* Cardiac pacemaker
* Expected survival time less than one year
* Expected poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-10-26 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Bladder cancer recurrence rate | 2 years
  Any bladder cancer recurrence at 2 years

SECONDARY OUTCOMES:
Progression of bladder cancer | 2 years
  Progression of bladder cancer in terms of T-category compared to the last resected tumour prior to randomisation
Mortality | 2 years
  Death due bladder cancer or other reasons
NMIBC24 quality of life questionnaire (QLQ) score | 2 years
  Side-effects related to the treatment measured with EORTC QLQ-NMIBC24
Adverse effects | 2 years
  Complications or adverse events related to bladder cancer or the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Boström, MD, PhD, Study Director — Turku University Hospital, Hospital District of Southwest Finland
Locations (7):
- Finland (7):
  - HYKS Peijas Hospital, Helsinki
  - Jyväskylä Central Hospital, Jyväskylä
  - Päijät-Häme Central hospital, Lahti
  - Mikkeli Central Hospital, Mikkeli
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pasin E, Josephson DY, Mitra AP, Cote RJ, Stein JP. Superficial bladder cancer: an update on etiology, molecular development, classification, and natural history. Rev Urol. 2008 Winter;10(1):31-43. PMID 18470273
- [Background] Sylvester RJ, van der Meijden AP, Oosterlinck W, Witjes JA, Bouffioux C, Denis L, Newling DW, Kurth K. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol. 2006 Mar;49(3):466-5; discussion 475-7. doi: 10.1016/j.eururo.2005.12.031. Epub 2006 Jan 17. PMID 16442208
- [Background] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Background] Prescott S, James K, Hargreave TB, Chisholm GD, Smyth JF. Radio-immunoassay detection of interferon-gamma in urine after intravesical Evans BCG therapy. J Urol. 1990 Nov;144(5):1248-51. doi: 10.1016/s0022-5347(17)39713-6. PMID 2122008
- [Background] Luo Y, Knudson MJ. Mycobacterium bovis bacillus Calmette-Guerin-induced macrophage cytotoxicity against bladder cancer cells. Clin Dev Immunol. 2010;2010:357591. doi: 10.1155/2010/357591. Epub 2010 Sep 1. PMID 20862387
- [Background] Brandau S, Riemensberger J, Jacobsen M, Kemp D, Zhao W, Zhao X, Jocham D, Ratliff TL, Bohle A. NK cells are essential for effective BCG immunotherapy. Int J Cancer. 2001 Jun 1;92(5):697-702. doi: 10.1002/1097-0215(20010601)92:53.0.co;2-z. PMID 11340575
- [Background] Morales A, Eidinger D, Bruce AW. Intracavitary Bacillus Calmette-Guerin in the treatment of superficial bladder tumors. J Urol. 1976 Aug;116(2):180-3. doi: 10.1016/s0022-5347(17)58737-6. PMID 820877
- [Background] Pan J, Liu M, Zhou X. Can intravesical bacillus Calmette-Guerin reduce recurrence in patients with non-muscle invasive bladder cancer? An update and cumulative meta-analysis. Front Med. 2014 Jun;8(2):241-9. doi: 10.1007/s11684-014-0328-0. Epub 2014 May 8. PMID 24810644
- [Background] Malmstrom PU, Sylvester RJ, Crawford DE, Friedrich M, Krege S, Rintala E, Solsona E, Di Stasi SM, Witjes JA. An individual patient data meta-analysis of the long-term outcome of randomised studies comparing intravesical mitomycin C versus bacillus Calmette-Guerin for non-muscle-invasive bladder cancer. Eur Urol. 2009 Aug;56(2):247-56. doi: 10.1016/j.eururo.2009.04.038. Epub 2009 Apr 24. PMID 19409692
- [Background] Chou R, Selph S, Buckley DI, Fu R, Griffin JC, Grusing S, Gore JL. Intravesical Therapy for the Treatment of Nonmuscle Invasive Bladder Cancer: A Systematic Review and Meta-Analysis. J Urol. 2017 May;197(5):1189-1199. doi: 10.1016/j.juro.2016.12.090. Epub 2016 Dec 24. PMID 28027868
- [Background] Sylvester RJ, van der MEIJDEN AP, Lamm DL. Intravesical bacillus Calmette-Guerin reduces the risk of progression in patients with superficial bladder cancer: a meta-analysis of the published results of randomized clinical trials. J Urol. 2002 Nov;168(5):1964-70. doi: 10.1016/S0022-5347(05)64273-5. PMID 12394686
- [Background] Bohle A, Bock PR. Intravesical bacille Calmette-Guerin versus mitomycin C in superficial bladder cancer: formal meta-analysis of comparative studies on tumor progression. Urology. 2004 Apr;63(4):682-6; discussion 686-7. doi: 10.1016/j.urology.2003.11.049. PMID 15072879
- [Background] Lamm DL, Blumenstein BA, Crissman JD, Montie JE, Gottesman JE, Lowe BA, Sarosdy MF, Bohl RD, Grossman HB, Beck TM, Leimert JT, Crawford ED. Maintenance bacillus Calmette-Guerin immunotherapy for recurrent TA, T1 and carcinoma in situ transitional cell carcinoma of the bladder: a randomized Southwest Oncology Group Study. J Urol. 2000 Apr;163(4):1124-9. PMID 10737480
- [Background] Di Stasi SM, Giannantoni A, Massoud R, Dolci S, Navarra P, Vespasiani G, Stephen RL. Electromotive versus passive diffusion of mitomycin C into human bladder wall: concentration-depth profiles studies. Cancer Res. 1999 Oct 1;59(19):4912-8. PMID 10519404
- [Background] Rajala P, Kaasinen E, Rintala E, Jauhiainen K, Nurmi M, Alfthan O, Lahde M. Cytostatic effect of different strains of Bacillus Calmette-Guerin on human bladder cancer cells in vitro alone and in combination with mitomycin C and interferon-alpha. Urol Res. 1992;20(3):215-7. doi: 10.1007/BF00299720. PMID 1615583
- [Background] Oosterlinck W, Kirkali Z, Sylvester R, da Silva FC, Busch C, Algaba F, Collette S, Bono A. Sequential intravesical chemoimmunotherapy with mitomycin C and bacillus Calmette-Guerin and with bacillus Calmette-Guerin alone in patients with carcinoma in situ of the urinary bladder: results of an EORTC genito-urinary group randomized phase 2 trial (30993). Eur Urol. 2011 Mar;59(3):438-46. doi: 10.1016/j.eururo.2010.11.038. Epub 2010 Dec 7. PMID 21156335
- [Background] Kaasinen E, Wijkstrom H, Malmstrom PU, Hellsten S, Duchek M, Mestad O, Rintala E; Nordic Urothelial Cancer Group. Alternating mitomycin C and BCG instillations versus BCG alone in treatment of carcinoma in situ of the urinary bladder: a nordic study. Eur Urol. 2003 Jun;43(6):637-45. doi: 10.1016/s0302-2838(03)00140-4. PMID 12767365
- [Background] Solsona E, Madero R, Chantada V, Fernandez JM, Zabala JA, Portillo JA, Alonso JM, Astobieta A, Unda M, Martinez-Pineiro L, Rabadan M, Ojea A, Rodriguez-Molina J, Beardo P, Muntanola P, Gomez M, Montesinos M, Martinez Pineiro JA; Members of Club Urologico Espanol de Tratamiento Oncologico. Sequential combination of mitomycin C plus bacillus Calmette-Guerin (BCG) is more effective but more toxic than BCG alone in patients with non-muscle-invasive bladder cancer in intermediate- and high-risk patients: final outcome of CUETO 93009, a randomized prospective trial. Eur Urol. 2015 Mar;67(3):508-16. doi: 10.1016/j.eururo.2014.09.026. Epub 2014 Oct 6. PMID 25301758
- [Background] Di Stasi SM, Giannantoni A, Stephen RL, Capelli G, Navarra P, Massoud R, Vespasiani G. Intravesical electromotive mitomycin C versus passive transport mitomycin C for high risk superficial bladder cancer: a prospective randomized study. J Urol. 2003 Sep;170(3):777-82. doi: 10.1097/01.ju.0000080568.91703.18. PMID 12913696
- [Result] Di Stasi SM, Giannantoni A, Giurioli A, Valenti M, Zampa G, Storti L, Attisani F, De Carolis A, Capelli G, Vespasiani G, Stephen RL. Sequential BCG and electromotive mitomycin versus BCG alone for high-risk superficial bladder cancer: a randomised controlled trial. Lancet Oncol. 2006 Jan;7(1):43-51. doi: 10.1016/S1470-2045(05)70472-1. PMID 16389183
- [Result] Gan C, Amery S, Chatterton K, Khan MS, Thomas K, O'Brien T. Sequential bacillus Calmette-Guerin/Electromotive Drug Administration of Mitomycin C as the Standard Intravesical Regimen in High Risk Nonmuscle Invasive Bladder Cancer: 2-Year Outcomes. J Urol. 2016 Jun;195(6):1697-703. doi: 10.1016/j.juro.2016.01.103. Epub 2016 Feb 2. PMID 26845426